CLINICAL TRIAL: NCT03338491
Title: Research Group RISKDYNAMICS, Sub-Project 8, Work Package 1, Study 2 (Student Sub-study): Addiction Risk: The Influence of Mindset Induction on the Effect of a Brief Intervention to Reduce Alcohol Use
Brief Title: Addiction Risk: Mindset Induction Effect on Brief Intervention
Acronym: AddRiskStud
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unexpected alcohol use increase identified in preliminary analysis after half of study enrollments
Sponsor: University of Konstanz (Other)
Responsible Party: Principal Investigator, Michael Odenwald, Director Outpatient Clinic or Psychotherapy, University of Konstanz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OD 113/2-1(3)
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Alcohol Drinking in College
MeSH Terms: conditions — Alcohol Drinking in College

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Induction of Implemental Mindset (Experimental): Psychological Intervention. Participants are asked to work on a brief paper-and-pencil task that has been shown to induce an Implemental Mindset according to the Mindset theory of action phases (Gollwitzer & Keller (2016). Mindset Theory. In: V. Zeigler-Hill, T.K. Shackelford (eds.), Encyclopedia of Personality and Individual Differences. New York: Springer).
  Interventions: Behavioral: Induction of Implemental Mindset
- Induction of Deliberative Mindset (Experimental): Psychological Intervention. Participants are asked to work on a brief paper-and-pencil task that has been shown to induce a Deliberative Mindset according to the Mindset theory of action phases (Gollwitzer & Keller (2016). Mindset Theory. In: V. Zeigler-Hill, T.K. Shackelford (eds.), Encyclopedia of Personality and Individual Differences. New York: Springer).
  Interventions: Behavioral: Induction of Deliberative Mindset
- Control (No Intervention): Participants will revive no induction of any mindset.

INTERVENTIONS:
Behavioral: Induction of Implemental Mindset — This induction of a psychological state was extensively studied in basic cognitive science. Gollwitzer & Keller (2016, p.3): "The implemental mindset is evoked by asking participants to think of a personal project for which they have already made the decision to act but did not initiate any action yet. Subsequently, participants are asked to list the steps necessary for successful goal attainment and to plan out in detail when, where, and how they intend to act on each of these steps."
  Arms: Induction of Implemental Mindset
Behavioral: Induction of Deliberative Mindset — This induction of a psychological state was extensively studied in basic cognitive science. Gollwitzer & Keller (2016, p.3): "The deliberative mindset is evoked by asking participants to (a) name an unresolved, important personal problem that is causing rumination but for which they have not made a decision yet and (b) reflect on whether to take action or not. Further, to enhance the depth of reflection, participants are requested to list a number of positive and negative, short- and long-term consequences of both deciding to act and deciding not to act; indicating the probability of the occurrence of each of these consequences is required."
  Arms: Induction of Deliberative Mindset

SUMMARY:
Brief Interventions (BI) based on Motivational Interviewing are effective to reduce alcohol use. In this study the investigators test the hypothesis that that an open Mindset increases the positive effects of BI.

University students take part in a voluntary screened for risky alcohol use. All students with risky alcohol use are eligible to the study and all receive the WHO's ASSIST-linked BI.

Participants receive a brief Mindset induction prior to receiving BI. They are are randomly assigned to either the induction of an open or a closed mindset according to the Mindset theory of action phases (Gollwitzer & Keller (2016). Mindset Theory. In: V. Zeigler-Hill, T.K. Shackelford (eds.), Encyclopedia of Personality and Individual Differences. New York: Springer).

The investigators measure the change in alcohol-related risk perception, treatment motivation and real alcohol drinking after the Brief Intervention in relation to the mindset induced before receiving the intervention.

ELIGIBILITY:
Inclusion Criteria:

* student status at University of Konstanz
* risky alcohol use in past 12 months

Exclusion Criteria:

* acute psychosis, acute suicidality, illiteracy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Questionnaire on Alcohol-related Risk Perception | 4 weeks
  Self-Report Measure that is filled out by the participant. This German questionnaire was developed by Klepper, Odenwald & Rockstroh (2016).
Alcohol Time-line Follow Back | 4 weeks
  Self-reported amount of standard alcohol units consumed. The assessment is made with the calendar method developed by Sobell & Sobell (1995)

SECONDARY OUTCOMES:
SOCRATES | 4 weeks
  Questionnaire: The Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES, Miller, W. R., & Tonigan, J. S. (1996). Assessing drinkers' motivation for change: The Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES). Psychology of Addictive Behaviors 10, 81-89.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Odenwald, PhD, Principal Investigator — University of Konstanz
Locations (1):
- University of Konstanz, Psychotherapy Outpatient Clinic, Konstanz, Germany

IPD SHARING:
Plan to Share IPD: Undecided